CLINICAL TRIAL: NCT01690559
Title: Ciprofloxacin Special Drug Use Investigation - To Investigate the Safety and Efficacy in Patients With Ciprofloxacin iv Administration Without Dilution
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Yakuhin, Ltd
Other Study IDs: 16516; CIPRO-IV-2010 (Other: company internal)
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Infection
Keywords: Ciprofloxacin; sepsis; infection; pneumonia; peritonitis; cholecystitis; cholangitis; anthrax
MeSH Terms: conditions — Infections; Sepsis; Pneumonia; Peritonitis; Cholecystitis; Cholangitis; Anthrax | interventions — Ciprofloxacin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patient treated with Ciproxan without dilution treatment in daily clinical practice
  Interventions: Drug: Cipro (Ciprofloxacin, BAYQ3939)

INTERVENTIONS:
Drug: Cipro (Ciprofloxacin, BAYQ3939) — Patient treated with Ciproxan without dilution treatment in daily clinical practice

SUMMARY:
This study is a post-marketing surveillance in Japan to investigate the safety especially focusing on injection site adverse events and efficacy in patients with Ciprofloxacin iv administration without dilution in the daily practice.It is a local prospective and observational study of patients who have received Ciproxan intravenously for sepsis, secondary skin infections followed by superficial burn, post-surgical or post-traumatic, pneumonia, peritonitis, cholecystitis, cholangitis, anthrax. A total of 500 patients are to be enrolled and assessed during the period of treatment with Ciproxan.

ELIGIBILITY:
Inclusion Criteria:

* - The mentioned bellow patients caused by the following bacteria which are sensitive to this drug: Indicated microorganisms:Staphylococcus, Enterococcus, Bacillus anthracis, Escherichia coli, Klebsiella , Enterobacter, Pseudomonas aeruginosa, Legionella. Indications: Sepsis, Secondary skin infections (superficial burn, operative wounds, trauma), Pneumonia, Peritonitis, Cholecystitis, Cholangitis, Anthrax
* The patients treated with this drug without dilution due to strict restriction of fluid intake.
* In hospitalized patients who retain consciousness ,and at the same time who are able to report (such as vascular pain) side effects..

Exclusion Criteria:

* Patients who are contraindicated based on the product label.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received Ciproxan iv administration without dilution in the daily practice among those with sepsis, secondary infection due to trauma, burn, or surgical wound, pneumonia, peritonitis, cholecystitis, cholangitis, and anthrax as the indications of this drug.
Sampling Method: Non-Probability Sample
Enrollment: 704 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) and serious adverse events (AEs) | After 8 days
Clinical efficacy by four grade (Response, Minor Response, No Response, and Indeterminable) at an investigator discretion | After 8 days

SECONDARY OUTCOMES:
ADR incidence rates classified by patient's background factors | After 8 days
Efficacy rate calculated with Response and Minor Response considered as responder | After 8 days
Efficacy rates classified by patient's background factors | After 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan